CLINICAL TRIAL: NCT05850481
Title: Role of Rotational Thromboelastometry and Platelet Indices as Predictors of Bleeding in Thrombocytopenic Patients.
Brief Title: Role of ROTEM and Platelet Indices in Thrombocytopenic Patients .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Abd Elazeem Saber Selim, Assistant Lecturer, Assiut University
Other Study IDs: ROTEM in thrombocytopenia
Record Dates: First submitted 2023-03-02; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Patients With Low Platelets Counts

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Investigate the role of thromboelastometry (ROTEM) parameters in the prediction of bleeding events in thrombocytopenic patients.
2. Interpretation of platelet indices in thrombocytopenic patients and detection of their role in prediction of bleeding in these patients .
3. Examine the correlations between ROTEM parameters, platelet indices in thrombocytopenic patients .

DETAILED DESCRIPTION:
Platelets are anucleate cells derived from megakaryocytes that play an important role in maintaining the integrity of the vascular endothelium and preventing haemorrhage. Adult platelet counts range from 150 - 450x10^3 / μL.The presence of a subnormal amount of platelets(<150 x 10^3 / μL)in circulating blood is referred to as thrombocytopenia, It is one of the most common haematological disorders and can become lifethreatening in case of severe disease. It could be due to a lack of platelet production or the degradation of platelets in the periphery. Hypoproliferative thrombocytopenias (aplastic anaemia, acute leukaemia) are one type of thrombocytopenia, while destructive thrombocytopenias (Idiopathic thrombocytopenia, secondry to SLE) are another. Bleeding is more likely in patients with severe thrombocytopenia.various reports have shown that platelet count is not a reliable predictor of clinically significant hemorrhage in thrombocytopenic patients Therefore, it may not be appropriate to use platelet count to guide treatment. Unfortunately, platelet function assays are often not sufficiently sensitive when platelet count is very low. As such, there remains the need to identify a predictor or set of parameters that can accurately assess the risk of hemorrhage in this patients.

The interpretation of platelet indices can aid in the initial care of thrombocytopenic patients ,Given the convenience and non-invasive nature of platelet indices calculation Although there are few studies in the literature on the significance of various platelet indices. the current study will be conducted to underline their importance in the diagnosis of thrombocytopenia.

Thromboelastography is a global coagulation test . The test is used to assess the change in elasticity over time of whole blood samples . Thromboelastography provides information about platelet function, coagulation, and fibrinolysis in just one assay monitoring.After improvement and automation, a thromboelastographic system known as ROTEM (rotational thromboelastometry) is now widely used in various clinical settings to determin the cause of bleeding in patients, evaluate bleeding risk, monitor the effect of anticoagulant drugs.and guide treatment.

The International Society on Thrombosis and Hemostasis (ISTH) is one of the well-known tools for bleeding assessment . The ISTH-BAT is a diagnostic questionnaire to screen patient depending on presence and absence of bleeding and also their severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thrombocytopenia and normal coagulation results
* Patients with and without significant bleeding events

Exclusion Criteria:

* patients with abnormal routine coagulation results (M3,liver diseases,........)
* patients who had received blood transfusions in the last 5 days.
* patients taking anticoagulant drugs or antiplatelet drugs .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients diagnosed as hypoproliferative thrombocytopenias(aplastic anaemia, acute leukaemia) and destructive thrombocytopenias (Idiopathic thrombocytopenia, secondry) with platelet count < 50 x 103 / μL and normal coagulation results
  * Patients with and without significant bleeding events
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
investigate the role of EXTEM in detection of bleeding risk in thrombocytopenic patients by using thromboelastometry (ROTEM) delta analyzer | baseline
  ROTEM assays will be performed using a ROTEM delta analyzer. Parameters such as EXTEM A10, EXTEM MCF, and EXTEM AUC will be obtained from EXTEM assay. This measurements will be used to predict risk of bleeding in patients with low platelet count
investigate the role of FIBTEM ROTEM parameter in detection of bleeding risk in thrombocytopenic patients by using thromboelastometry (ROTEM) delta analyzer | baseline
  FIBTEM ROTEM parameter will be performed using a ROTEM delta analyzer Platelet MCE will be calculated by subtracting FIBTEM MCE from EXTEM MCE (Platelet MCE = EXTEM MCE - FibTEM MCE).This measurements will be used to predict risk of bleeding in patients with low platelet count

SECONDARY OUTCOMES:
Measuring of Platelet distribution width (%) | baseline
  Interpretation the role of Platelet parameter (Platelet distribution width (%) )and detection of their role in prediction of bleeding in patients with low platelet count
Measuring of Mean platelet volume (fL). | baseline
  Interpretation the role of Platelet parameters (Mean platelet volume (fL)). and detection of their role in prediction of bleeding in these patients

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mohamed Helbawi, Lecturer, Study Director — Clinical pathology department ,Assiut University Hospital; Mohammed Ashraf Mahmoud, Lecturer, Study Director — Clinical pathology department ,Assiut University Hospital

REFERENCES:
- [Background] Parise LV. Introduction to a review series: megakaryocytes to platelets in health and disease. Blood. 2016 Mar 10;127(10):1215. doi: 10.1182/blood-2015-11-664029. Epub 2016 Jan 19. No abstract available. PMID 26787732
- [Background] Middelburg RA, Carbaat-Ham JC, Hesam H, Ragusi MA, Zwaginga JJ. Platelet function in adult ITP patients can be either increased or decreased, compared to healthy controls, and is associated with bleeding risk. Hematology. 2016 Oct;21(9):549-51. doi: 10.1080/10245332.2016.1180097. Epub 2016 May 9. PMID 27159138
- [Background] Nguyen TH, Tran TT, Hoang TT, Nguyen TT. Rotational thromboelastometry parameters as predicting factors for bleeding in immune thrombocytopenic purpura. Hematol Oncol Stem Cell Ther. 2021 Mar;14(1):27-32. doi: 10.1016/j.hemonc.2020.05.003. Epub 2020 May 15. PMID 32446931
- [Background] Ni L, Xue P, An C, Yu X, Qu J, Yao Y, Li Y. Establishment of Normal Range for Thromboelastography in Healthy Middle-Aged and Elderly People of Weihai in China. J Healthc Eng. 2021 Nov 28;2021:7119779. doi: 10.1155/2021/7119779. eCollection 2021. PMID 34876966
- [Background] Saqlain N, Fateen T, Tufail H, Mazher N. Utility of the ISTH bleeding assessment tool (BAT) in diagnosis of Glanzmann Thrombasthenia patients. Pak J Med Sci. 2022 Mar-Apr;38(4Part-II):791-795. doi: 10.12669/pjms.38.4.5361. PMID 35634602